CLINICAL TRIAL: NCT04236427
Title: Efficacy and Safety of Chinese Medicine Angong Niuhuang Wan for the Treatment of the Stroke: A Randomized, Double-blind,Placebo Controlled Clinical Trial
Brief Title: Efficacy and Safety of Angong Niuhuang Wan for Stroke
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Alexander Lau, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ANP study
Record Dates: First submitted 2019-10-14; First posted 2020-01-22 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Stroke (CVA) or TIA
MeSH Terms: conditions — Stroke | interventions — Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Chinese Medicine of Angong Niuhuang Wan
  Interventions: Drug: Angong Niuhuang Wan
- Placebo Group (Placebo Comparator): Placebo of Angong Niuhuang Wan
  Interventions: Drug: Angong Niuhuang Wan Placebo

INTERVENTIONS:
Drug: Angong Niuhuang Wan — Angong Niuhuang Wan 3g
  Other Names: Active drug
  Arms: Treatment Group
Drug: Angong Niuhuang Wan Placebo — Angong Niuhuang Wan Placebo 3g
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
To evaluate the efficacy and safety of using Chinese Medicine Angong Niuhuang Wan in stroke patients, the modified Rankin Scale (mRS) score will be used as primary outcome, the National Institutes of Health Stroke Scale (NIHSS) score, The Modified Barthel Index (MBI) score and the Montreal Cognitive Assessment (MoCA) scores will be used as secondary outcome measures.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled trial which is used to further determine the effectiveness of Angong Niuhuang Wan in treating stroke patients on top of the standard conventional treatment, also to evaluate the improvement level on quality of life of post-stroke after using Angong Niuhuang Wan. The effect of Angong Niuhuang Wan on liver and kidney function will be focused and using NMR techniques to analysis metabolomics to further study the safety and effectiveness of Angong Niuhuang Wan on the prevention and treatment of stroke.

It is a 24-week trial, Double-blind treatment for 1 week, follow up visit for 23 weeks. All participant will have study blood taking for renal and liver function test and questionnaires assessment during study visits. Informed consent will be obtained before study enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults aged 40 or above;
2. diagnosed as a stroke by a neurologist, with imaging of CT or MRI support;
3. Neurologist confirms the symptoms of stroke occur within 28 days and are clinically stable. In the past 48 hours, the condition of the nervous system has not deteriorated significantly;
4. TCM diagnosis is a stroke and belongs to a heat syndrome;
5. There is a movement defect caused by stroke;
6. The severity of stroke was scored 5-25 by the National Institutes of Health Brain Stroke Scale (NIHSS);
7. Informed consent will be given by participant or its representatives

Exclusion Criteria:

1. The movement defects are not associated with stroke. Before commencement of study treatment, patient has physical activity dysfunction caused by lameness , osteoarthritis, rheumatoid arthritis, gouty arthritis, etc. that may affect neurological function examination;
2. Subjects are unlikely to come back for follow-up visits during the 24-week study period;
3. The subject has a brain tumor on a computed tomography scan (CT);
4. The subject has thrombocytopenia (known platelet count <100,000 / mm3) or coagulopathy disease;
5. Taking warfarin or other anticoagulant;
6. Concomitant diseases such as severe hypertension or diabetes;
7. Comorbidities or complications associated with drug evaluation;
8. Pregnant or breast-feeding female.
9. The alanine aminotransferase (ALT) value is 1.5 times higher than the normal maximum value in liver function test and the estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m2 in the renal function test.
10. Present the sign of pure yin syndrome or yin / yang defecation in TCM diagnosis;
11. Subject has G6PD
12. Known swallowing problem
13. Dependent in all daily life activities

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Score of neurological deficit and adverse events | 24 weeks
  compare the therapeutic effects, the score of neurological deficit and adverse events between the two groups by using questionnaire of mRS, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Mortality and recurrence rates of stroke | 24 weeks
  Compare the mortality and recurrence rates of stroke between two groups also the abilities of daily ability using questionnaires of NIHSS (higher scores mean a worse outcome), mBI and MOCA-HK (higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Yuk-lun LAU, Post-doc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No